CLINICAL TRIAL: NCT06418035
Title: Acquisition of Daily Living Skills in Autistic Children: Comparison Between Video-modeling Mediated by iPad (QR Code) and Modeling With a Human Operator
Brief Title: Acquisition of Daily Living Skills in Autistic Children: Comparison Between QR Code and a Human Operator
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Messina, Italy (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2024-005
Record Dates: First submitted 2024-05-02; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: autism; children; technology; daily living skills; video modeling; applied behavior analysis
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: treatment with technological tool (Experimental): The intervention will be structured according to Applied Behavioral Analysis. The target activities to be performed are shown on the iPad through video-modeling. The child, using iPad, scans QR codes placed in various stations of the HomeLab, near the place where the target autonomy will be carried out. HomeLab is a room that simulates a real apartment with various domestic areas and allows the child to feel as comfortable as at home.
  Interventions: Behavioral: Video modeling by scanning Qr code
- Control group: traditional treatment without technological tool (Other): The intervention will be structured according to Applied Behavioral Analysis. The target activities to be performed within HomeLab are shown, live, by an operator who acts as a model.
  Interventions: Behavioral: Modeling traditional method

INTERVENTIONS:
Behavioral: Video modeling by scanning Qr code — The protocol activity carried out by the experimental group will involve the use of the QR Code: in the operator's presence, the child scans the code through a technological device and watches the video of the activity to be played later in the HomeLab.
  Arms: Experimental group: treatment with technological tool
Behavioral: Modeling traditional method — The control group will carry out the protocol activities in a traditional way, without technological tools. The child observes the operator who shows the live activity inside the HomeLab.
  Arms: Control group: traditional treatment without technological tool

SUMMARY:
Autism spectrum disorder (ASD), is a condition characterized by deficits in social communication and mutual interaction, as well as repetitive and restricted behaviors and interests. This condition manifests itself differently in each individual and can vary greatly in severity and impact on daily life.

Autistic children may present various challenges and difficulties in developing daily living skills (DLS). These difficulties may relate to various areas, such as personal autonomy and domestic autonomy. For example, they may have difficulties in acquiring personal hygiene skills, such as dressing and tying their shoes independently. They may have difficulty performing household tasks, such as setting the table, preparing a simple meal, or folding a t-shirt. These difficulties may require specific support and training to help autistic children develop personal autonomy skills and achieve greater independence in different areas of their daily lives. Improving and developing DLS is an important goal in order to improve the quality of life and independence of children with autistic conditions.

This protocol aims to acquire new useful DLS within the various settings of daily life. The hypothesis of the present study is the following: video modeling, through the use of the iPad (Qr code scanning), can be more effective in promoting autonomy in children with ASD, compared to a control group that receives a traditional training, without the use of technological instrumentation.

DETAILED DESCRIPTION:
In this study, participants will be randomly assigned to an experimental or control group.

Both groups will be subjected to applied behavior analysis (ABA) procedures: the behavioral procedure, called modeling, is a technique in which the participant observes and imitates a target behavior of a operator who serves as a "model." Such modeling can be in vivo or remotely (via video).

Also included is the use of task analysis with the aim of identifying all the smaller teachable units of a complex behavior, the sub-targets, that make up a behavioral chain. The participant, after observing the entire target task performed by the model, in turn performs the behavioral chain.

Based on the data collected at baseline, the operator will deliver a simultaneous response prompt to promote errorless learning only in the individual subtasks absent in the participant's repertoire. The mode in which prompts will be delivered will be of the "least to most" type, that is, from least to most intrusive help, according to the following hierarchy:

P1. gestural prompt P2. verbal-vocal prompt P3. total physical prompt The operator will begin by delivering the least intrusive prompt, P1 (gestural). If the participant does not deliver the correct behavior within 5'', the operator will move to the next most intrusive prompt, P2 (verbal-vocal); if the participant does not deliver the correct behavior within 5'', the operator will move to the next most intrusive prompt, P3 (total physical).

Both groups will be subjected to n° 5 personal autonomies, during every experimental sessions.

The experimental group, inside the HomeLab, will scan the Qr code using iPad and view the video-modeling of the target activity to be performed; the control group will carry out the target activity, inside the HomeLab, in a traditional way, without technological instrumentation and will observe the operator who acts as a model live.

This experimental study will be implemented for a total of 6 months with biweekly frequency lasting 45 minutes per session. At the end of each session, the percentage of independent correct answers will be calculated. The acquisition criterion for defining "acquired" target autonomy is the achievement of 90% independent responses for 3 consecutive sessions.

Families of children with ASD will be recruited from the Institute for Biomedical Research and Innovation of the Italian National Research Council (IRIB-CNR) in Messina, Italy.

Eligible participants who meet the inclusion criteria will receive written information about the procedure and will be asked to sign the informed consent form indicating their willingness to participate in the study. Only those individuals who have provided informed consent will be randomly assigned to the experimental or control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder;
* IQ below 80 assessed by means of WISC IV or Leiter-3;
* Passing the ABLLS-R "imitation" and "visual performance" tests

Exclusion Criteria:

* Presence of other medical disorders;
* Absence of imitative and visual-perceptual skills.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
WISC-IV (Wechsler Intelligence Scale for Children-4° edition) | The evaluation session will be scheduled pre-intervention (T0). The test needs approximately 65-80 minutes to complete.
  Wechsler Intelligence Scale for Children Fourth edition (WISC-IV) is a clinical tool for assessing the cognitive abilities of children and young people between the ages of 6 years and 16 years and 11 months.
  The WISC-IV scales are as follows:
  index of verbal comprehension (ICV), range weighted scores (min 46 - max154); index visuoperceptual reasoning (IRP), range weighted scores (min 41- max 159); index working memory (IML) range weighted scores (min 46 - max 154); processing speed index (IVE) range weighted scores (min 47 - max 153); intelligence quotient IQ (min 40 - max 160). For each sub-scale higher score corresponds to better performance.
Griffiths Mental Development Scales (GMDS-3rd) | The evaluation session will be scheduled pre-intervention (T0). Test administration is individual and lasts about 90 minutes.
  The Griffiths III are an instrument for assessing child development from birth to 6 years of age. The Griffiths III are based on an integrated model of development, conceived as consisting of various domains that interact and influence each other and determine the child's development.
  Scale A. Basics of learning, range scores (min 0 - max 20) Scale B. Language and communication, range scores (min 0 - max 20). Scale C. Oculo-manual coordination, range scores (min 0 - max 20) Scale D. Personal-social-emotional, range scores (min 0 - max 20) Scale E. Gross-motor, range scores (min 0 - max 20) For each sub-scale higher score corresponds to better performance. The Griffiths III enables information to be obtained about each area of development considered (each scale can also be used individually), to draw a developmental profile in terms of strengths and weaknesses, but also to have an indication of the child's overall level of development.
Vineland Adaptive Behavior Scales-II (Vineland-II) | The tests will be scheduled pre intervention (T0) and at the study conclusion, at 6 months (T1).The T0 and T1 evaluations were conducted to determine whether the protocol carried out made a change. The test needs about 60 minutes.
  The Vineland-II, a revision of the Vineland Adaptive Behavior Scales, assess adaptive behavior (AB), i.e., the activities that the individual habitually performs to meet the expectations of personal autonomy and social responsibility characteristic of people of the same age and cultural background.
  Specifically, they aim to measure AB in the domains Communication, range scores (min 0 -max 160), Skills of Daily Living, range scores (min 0 - max 160) Socialization, range scores (min 0- max 160) (in individuals from 0 to 90 years of age) and Motor Skills, range scores (min 0 -max 160) (in individuals from 0 to 7 years of age and 56 to 90 years of age). For each sub-scale higher score corresponds to better performance.
  Assessment of AB is necessary for diagnosis of intellectual disability disorder and, in accordance with DSM-5, for assessment of the level of severity of the disorder.
  The Vineland-IIs consist of 4 scales divided into 11 subscales. They also provide an overall AB index.
The Assessment of Basic Language and Learning Skills-Revised (ABLLS-R) | The tests will be scheduled pre intervention (T0) and at the study conclusion, at 6 months (T1). The administration time is approximately 60 minutes.
  The Assessment of Basic Language and Learning Skills- Revised (ABLLS-R) is tracking system based on the basic language and functional skills of an individual with autism and other developmental delays. It is used as a tool to help develop individualized curricula to teach language and other critical skills to children with autism or other developmental disabilities. The ABLLS-R focuses on 25 skills in the areas of language, social interaction, self-help, academic and motor skills. The evaluation of this tool helps to identify the skills necessary for the child to communicate effectively and to identify obstacles that prevent the child from acquiring new skills. For research purposes, the evaluation will focus on self-help skills, specifically: Dressing Skills (min 0 - max 30), Feeding-related autonomies ( min 0 - max 20) Personal care skills ( min 0 - max 14), Toileting Skills ( min 0 max 20). For each sub-scale higher score corresponds to better performance.
Psychoeducational profile-3 (Pep-3) | The questionnaire will be scheduled pre intervention (T0) and at the study conclusion, at 6 months (T1). The administration time of the questionnaire for parents is 45 minutes.
  PEP-3 assesses learning inhomogeneity, strengths and weaknesses, and related developmental disabilities in children with autism and pervasive developmental disorders and children with developmental difficulties that are difficult to test (age range 2 to 12 years).
  It is part of the TEACCH materials for individualized psychoeducational assessment and intervention for children with Autism Spectrum Disorder.
  The test consists of two main components:
  1. The Performance section (10 subtests)
  2. The questionnaire for parents (3 subtest). For the purpose of the research, only the parental questionnaire will be used. It investigates: problem behavior range scores (min 1 - max 20.) , personal autonomy range scores (min 1 - max 20.), adaptive behavior range scores (min 1 - max 20.).
  For each sub-scale higher score corresponds to better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR)
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mclay, Laurie & Carnett, Amarie & van der Meer, Larah & Lang, Russell. (2015). Using a Video Modeling-Based Intervention Package to Toilet Train Two Children with Autism. Journal of Developmental and Physical Disabilities. 27. 10.1007/s10882-015-9426-4.
- [Background] Drysdale, Bradley & Lee, Clara & Anderson, Angelika & Moore, Dennis. (2014). Using Video Modeling Incorporating Animation to Teach Toileting to Two Children with Autism Spectrum Disorder. Journal of Developmental and Physical Disabilities. 27. 10.1007/s10882-014-9405-1.
- [Background] Popple B, Wall C, Flink L, Powell K, Discepolo K, Keck D, Mademtzi M, Volkmar F, Shic F. Brief Report: Remotely Delivered Video Modeling for Improving Oral Hygiene in Children with ASD: A Pilot Study. J Autism Dev Disord. 2016 Aug;46(8):2791-2796. doi: 10.1007/s10803-016-2795-4. PMID 27106570
- [Background] Lee, Clara & Anderson, Angelika & Moore, Dennis. (2014). Using Video Modeling to Toilet Train a Child with Autism. Journal of Developmental and Physical Disabilities. 26. 10.1007/s10882-013-9348-y.